CLINICAL TRIAL: NCT06891404
Title: The Relationship Between Nurse-Led Health Belief Model-Based Education and Genital Hygiene Behaviors and Attitudes Toward the Prevention of Urinary Tract Infections
Brief Title: The Relationship Between Nurse-Led Health Belief Model-Based Education and Genital Hygiene and UTI Prevention Attitudes
Acronym: Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Merve Kolcu, Assistant professor, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2025/03
Record Dates: First submitted 2025-03-17; First posted 2025-03-24 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Health Belief Model; Education
Keywords: Health Belief Model; Education; Genital hygiene; Infections
MeSH Terms: conditions — Infections

STUDY DESIGN:
Intervention Model Description: The study will be conducted with 122 students, 61 controls and 61 interventions.
Who Masked: Participant
Masking Description: 2
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): The study will involve female students aged 18-49 who are studying at the Faculty of Health Sciences of a private university. Data will be collected via a pre-structured form using Google Forms. A pre-test will be applied to the students, followed by Health Belief Model (HBM)-based Genital Hygiene Education. The objectives of the education will be prepared in line with the sub-dimensions of the HBM, such as perceived susceptibility, perceived severity, perceived benefits, perceived barriers, self-efficacy, and cues to action. The education is planned to last a total of 4 class hours (160 minutes). The education will be conducted face-to-face in a classroom setting.Two weeks after the training, the students' behaviors and attitudes will be evaluated using the prepared data collection tool.
  Interventions: Other: Nurse-Led Health Belief Model-Based Education
- Control (No Intervention): The study will involve female students aged 18-49 who are studying at the Faculty of Health Sciences of a private university. Data will be collected via a pre-structured form using Google Forms. This group will not receive any education, but after the intervention group completes the education, a post-test will be conducted with this group as well.

INTERVENTIONS:
Other: Nurse-Led Health Belief Model-Based Education — Topic of the Training:
  Importance of Genital Hygiene Behaviors Definition of Urinary Tract Infection (UTI) Complications that may arise if left untreated Effects on daily life Proper toilet hygiene Selection and cleaning of underwear Menstrual hygiene Importance of sexual hygiene Common Misconceptions About Genital Hygiene Behaviors
  Arms: Experimental

SUMMARY:
Objective: This study seeks to enhance the hygiene awareness of students receiving education in the healthcare field, contributing to the development of healthy lifestyle habits. Additionally, the study's findings will provide essential data for improving educational programs and establishing strategies for protecting urogenital health.

Materials and Methods: The data for the study will be collected using the Descriptive Characteristics Form, the Genital Hygiene Behaviors Scale, and the Health Belief Scale for the Prevention of Urinary Tract Infections. The data analysis will be conducted using the Statistical Package for Social Sciences (SPSS) 25.0 Windows program, with a significance level of p<0.05 considered statistically significant. The normality distribution of the data will be examined, and Cronbach's Alpha internal consistency analysis will be performed to assess the validity and reliability of the scales. For the analysis of descriptive data, mean, standard deviation, frequency, and percentage will be used. The comparison of ordinal measurements will be analyzed using the paired t-test for repeated measures in dependent groups.

Design: Randomized controlled.

The population of the study will consist of students enrolled in the Departments of Child Development, Nutrition and Dietetics, Health Management, and Social Work at the Faculty of Health Sciences of a private university. Using the G*Power program, with 1-β = 0.95 power, α = 0.05 error level, and an effect size of f = 0.6, the sample size was determined to be 122 students (61 in the intervention group and 61 in the control group).

DETAILED DESCRIPTION:
Genital hygiene is one of the fundamental health behaviors that play a crucial role in protecting women's reproductive health. The reproductive age, defined as 15-49 years, is the period in which reproductive health issues are most frequently observed. It is reported that approximately one million women worldwide experience genital infections each year, and 75% of women have a history of vaginal infection. In developing countries, this issue is a significant public health concern that women encounter at least once in their lifetime. In Turkey, regional studies indicate that both genital infections and risky hygiene behaviors that may lead to vaginal infections are prevalent. Especially among young women, adopting proper hygiene habits is crucial in preventing genital infections, urinary tract infections (UTIs), and other urogenital health problems.

The Health Belief Model (HBM) is a widely used theoretical framework for understanding and improving individuals' health behaviors. HBM aims to explain individuals' perceptions of a disease or health problem and how these perceptions influence their behaviors. This model consists of several components: perceived susceptibility, perceived severity, perceived benefits, perceived barriers, self-efficacy, and cues to action. Educational programs are expected to increase individuals' awareness based on these components and promote positive behavioral changes in hygiene practices.

Hygiene education plays a vital role in maintaining genital hygiene. Various studies in the literature examine the relationship between education and young women's urogenital health. Research findings indicate that female students have knowledge gaps and that students who receive genital hygiene education adopt more conscious hygiene practices. However, experimental studies investigating the effect of HBM-based genital hygiene education on genital hygiene behaviors and attitudes toward the prevention of urinary tract infections remain limited.

In this context, the present study aims to evaluate the relationship between nurse-led HBM-based education provided to students of the Faculty of Health Sciences and their genital hygiene behaviors and attitudes toward UTI prevention.

This study seeks to enhance the hygiene awareness of students receiving education in the healthcare field, contributing to the development of healthy lifestyle habits. Additionally, the study's findings will provide essential data for improving educational programs and establishing strategies for protecting urogenital health.

ELIGIBILITY:
Inclusion Criteria:

* To agree to participate in the study, to fully attend the scheduled training

Exclusion Criteria:

* Refusing to participate in the study,
* having previously taken a course on women's reproductive health and genital hygiene,
* incomplete attendance at the training,
* incomplete filling out of the data collection tool.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 122 (Actual)
Dates: Start 2025-03-16 (Actual); Primary Completion 2025-06-15 (Actual); Study Completion 2025-08-15 (Actual)

PRIMARY OUTCOMES:
The Descriptive Characteristics Form | 5 minutes
  Consists of 14 items prepared by the researchers based on the literature.

SECONDARY OUTCOMES:
Genital Hygiene Behavior Scale | 15 minute
  The GHBS was developed to assess women's genital hygiene behaviors and consists of 23 items rated on a 5-point Likert scale (Karahan, 2017). The scale includes three subdimensions: "General Hygiene Practices" (items 1-12), "Menstrual Hygiene" (items 13-20), and "Awareness of Abnormal Symptoms" (items 21-23). Items are scored from 5 ("strongly agree") to 1 ("strongly disagree"), with items 7, 14, 19, 20, and 23 reverse coded. The total score ranges from 23 to 115, with higher scores indicating more positive genital hygiene behaviors.
Health Belief Scale for the Prevention of Urinary Tract Infections | 15 minute
  The HBS-UTI was developed to evaluate women's health beliefs regarding the prevention of urinary tract infections within the framework of the Health Belief Model (Kaçar & Kolaç, 2024). The scale comprises 26 items rated on a 5-point Likert scale and includes six subdimensions: "perceived benefit", "perceived obstacle", "perceived seriousness", "perceived sensitivity", "health motivation" and "self-efficacy". Possible scores range from 26 to 130, with higher scores reflecting stronger health beliefs toward the prevention of UTIs. The original Cronbach's alpha coefficient was 0.88, and in the present study it was calculated as 0.91.

CONTACTS AND LOCATIONS:
Overall Officials: Merve KOLCU, PhD, Principal Investigator — merve.kolcu@sbu.edu.tr; Nur Bahar KURU AKTURK, Msc, Study Chair — nurbaharkuru@arel.edu.tr; Aydan YILMAZ, Msc, Study Chair — aydan.yilmaz@sbu.edu.tr; Beyzanur ISBAY AYDEMIR, PhD(c), Study Chair — beyzanurisbay@aydin.edu.tr
Locations (1):
- University of Health Sciences, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No